CLINICAL TRIAL: NCT00466726
Title: Phase II Multicenter Study of P210-B3A2 Derived Peptide Vaccine in Chronic Myeloid Leukemia Patients in Complete Cytogenetic Response With Persistent Molecular Residual Disease During Imatinib Treatment
Brief Title: Vaccine Therapy in Treating Patients With Philadelphia Chromosome-Positive Chronic Myelogenous Leukemia
Acronym: CML0206
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CML 0206; 2006-006189-40 (EudraCT Number); NCT00452933 (obsolete NCT alias)
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Results first posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Leukemia
Keywords: chronic myelogenous leukemia, BCR-ABL1 positive; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase | interventions — sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: bcr-abl p210-b3a2 breakpoint-derived multipeptide vaccine
Biological: sargramostim

SUMMARY:
RATIONALE: Vaccines made from peptides may help the body build an effective immune response to kill cancer cells. Colony-stimulating factors, such as GM-CSF, may increase the number of immune cells found in bone marrow or peripheral blood. Giving booster vaccinations may make a stronger immune response and prevent or delay the recurrence of cancer.

PURPOSE: This phase II trial is studying how well vaccine therapy works in treating patients with Philadelphia chromosome-positive chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the activity of bcr-abl p210-b3a2 breakpoint-derived pentapeptide vaccine (CMLVAX100), in terms of peripheral blood bcr-abl/abl ratio reduction, in patients with Philadelphia chromosome-positive chronic myelogenous leukemia.

Secondary

* Determine the reduction of molecular residual disease at 3 months in patients treated with this vaccine.
* Determine the reduction of molecular residual disease at 12 months in patients treated with maintenance boosts of this vaccine.
* Determine the rate of complete molecular response at any time after vaccination.
* Determine in vivo and in vitro peptide-specific immune response induced by the vaccine.

OUTLINE: This is a prospective, nonrandomized, open-label, multicenter study.

Patients receive sargramostim (GM-CSF) subcutaneously (SC) on days 1 and 2 and bcr-abl p210-b3a2 breakpoint-derived pentapeptide vaccine (CMLVAX100) SC on day 2. Treatment repeats every 2 weeks for 6 courses. Patients then receive CMLVAX100 SC once monthly for 3 months and then once every 3 months for 6 months (for a total of 1 year). Patients may receive additional CMLVAX100 SC every 6 months for at least 3 years. Treatment continues in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 69 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic myelogenous leukemia (CML) meeting the following criteria:

  * Philadelphia chromosome positive disease
  * b3a2 breakpoint mutation
* Prior treatment with conventional imatinib mesylate for ≥ 18 months required

  * Complete cytogenetic response documented on ≥ 2 different examinations

    * Persistence of molecularly detectable residual disease (any level of bcr-abl transcript)
  * Patients continue to receive imatinib mesylate at the same dose (conventional treatment) during study treatment

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Bilirubin ≤ 2 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No severe active infection or other serious medical illness that would preclude study completion
* No known immunodeficiency
* No autoimmune disorders

PRIOR CONCURRENT THERAPY:

* No concurrent immunosuppression or systemic immunosuppressive medication
* No concurrent dose escalation of imatinib mesylate
* No other concurrent investigational products

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2007-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Bocchia, MD, Study Chair — Nouvo Policlinico "LE SCOTTE'
Locations (17):
- Italy (17):
  - Universita Degli Studi di Bari, Bari
  - Ospedali Riuniti di Bergamo, Bergamo
  - Istituto di Ematologia "Lorenzo e A. Seragnoli" - Università degli Studi di Bologna - Policlinico S. Orsola - Malpighi, Bologna
  - USD Trapianti di midollo per adulti - Cattedra di Ematologia - Università degli Studi di Brescia, Brescia
  - Università di Catania - Cattedra di Ematologia - Ospedale 'Ferrarotto', Catania
  - Ospedale Regionale A. Pugliese, Catanzaro
  - Federico II University Medical School, Naples
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - Azienda Ospedale S. Luigi at University of Torino, Orbassano
  - spedali Riuniti "Villa Sofia-Cervello", Palermo
  - Ospedale Sant' Eugenio, Rome
  - Universita Degli Studi "La Sapeinza", Rome
  - Policlinico A. Gemelli - Universita Cattolica del Sacro Cuore, Rome
  - Unità Operativa di Oncologia - Presidio Ospedaliero N. Giannetasio - Azienda ASL 3, Rossano
  - Ematologia - Dipartimento di Medicina Clinica e Sperimentale, Sassari
  - Nouvo Policlinico "LE SCOTTE', Siena
  - Policlinico Universitario Udine, Udine

REFERENCES:
- [Result] BCR-ABL Derived Peptide Vaccine in Chronic Myeloid Leukemia Patients with Molecular Minimal Residual Disease During Imatinib: Interim Analysis of a Phase 2 Multicenter GIMEMA CML Working Party Trial.
- See also: GIMEMA Foundation website — http://www.gimema.it

RESULTS

PARTICIPANT FLOW:
Groups:
- Chronic Myeloid Leukemia (CML) Patients: Study population
Period: Overall Study
Arm/Group | Chronic Myeloid Leukemia (CML) Patients
Started | 57
Completed | 43
Not Completed | 14
Not completed — Not evaluable for response | 14

BASELINE CHARACTERISTICS:
Arm/Group | Chronic Myeloid Leukemia (CML) Patients
Number analyzed (Participants) | 43
Age, Continuous [Median (Full Range); unit: years] | 56.5 [29 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Showing a Reduction by at Least 50% of Peripheral Blood BCR-ABL/ABL Ratio Compared to the Individual Prevaccine Level
Description: Response rate evaluated after immunization and reinforcement boosts (evaluation after 6 months, ) and persisting at the 9th month (after 10th vaccination)
Time Frame: At 6 and 9 months
Measure: Number; unit: participants
Arm/Group | Chronic Myeloid Leukemia (CML) Patients
Number analyzed (Participants) | 43
participants
  50% reduction at 6 months | 22
  50% reduction at 9 months | 14

2. Secondary Outcome: Number of Patients With Undetectable Transcript at Any Time After Immunization
Time Frame: Up to 6 months
Measure: Number; unit: participants
Arm/Group | Chronic Myeloid Leukemia (CML) Patients
Number analyzed (Participants) | 43
participants | 14

3. Secondary Outcome: Number of Patients With Peptide-specific Immune Response Induced by the Vaccinations
Description: A significant in vitro b3a2-peptide-specific CD4+ T cell proliferation
Time Frame: At 9 months
Measure: Number; unit: participants
Arm/Group | Chronic Myeloid Leukemia (CML) Patients
Number analyzed (Participants) | 43
participants | 29

ADVERSE EVENTS:
Arm/Group | Chronic Myeloid Leukemia (CML) Patients
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 4/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Myeloid Leukemia (CML) Patients (N=43)
Mild fever (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No